CLINICAL TRIAL: NCT02556203
Title: Global Multicenter, Open-label, Randomized, Event-driven, Active-controlled Study Comparing a rivAroxaban-based Antithrombotic Strategy to an antipLatelet-based Strategy After Transcatheter aortIc vaLve rEplacement (TAVR) to Optimize Clinical Outcomes
Brief Title: Global Study Comparing a rivAroxaban-based Antithrombotic Strategy to an antipLatelet-based Strategy After Transcatheter aortIc vaLve rEplacement to Optimize Clinical Outcomes
Acronym: GALILEO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Imbalance in the efficacy and safety endpoints between treatment arms in favor of comparator
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17938; 2015-001975-30 (EudraCT Number)
Record Dates: First submitted 2015-09-05; First posted 2015-09-22 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Transcatheter Aortic Valve Replacement
Keywords: TAVR; TAVI; Transfemoral aortic valve implantation
MeSH Terms: interventions — Rivaroxaban; Aspirin; Clopidogrel; acarboxyprothrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Xarelto, BAY59-7939) (Experimental): Subjects were treated with Rivaroxaban (10mg once-daily) and ASA (75-100mg once-daily) within first 90 days after randomization. After 90 days, ASA was discontinued and rivaroxaban (10mg once-daily) was to be continued alone. In the event of NOAF (New Onset of Atrial Fibrillation), subjects should be switched to rivaroxaban (20/15mg once-daily) and ASA (75-100mg once-daily) within first 90 days. After 90 days, ASA was discontinued and rivaroxaban (20/15mg once-daily) was to be continued alone.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Acetylsalicylic Acid (ASA)
- Antiplatelet (Active Comparator): Subjects were treated with clopidogrel (75mg once-daily) and ASA (75-100mg once-daily) within first 90 days after randomization. After 90 days, clopidogrel was discontinued and ASA (75-100mg once-daily) was to be continued alone. In the event of NOAF, subjects should start treatment of open-label VKA to target INR 2 to 3 (according to guidelines) and ASA (75-100mg once-daily) within first 90 days. After 90 days, ASA was discontinued and VKA was to be continued alone.
  Interventions: Drug: Acetylsalicylic Acid (ASA); Drug: Clopidogrel; Drug: Vitamin K antagonist (VKA)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 10mg OD (once-daily)
  Arms: Rivaroxaban (Xarelto, BAY59-7939)
Drug: Acetylsalicylic Acid (ASA) — 75-100mg OD
Drug: Clopidogrel — 75mg OD
  Arms: Antiplatelet
Drug: Rivaroxaban (Xarelto, BAY59-7939) — In case of NOAF, 20/15 mg OD (once-daily)
  Arms: Rivaroxaban (Xarelto, BAY59-7939)
Drug: Vitamin K antagonist (VKA) — In case of NOAF, Open-label VKA therapy to target international normalized ratio (INR) 2-3, according to guidelines
  Arms: Antiplatelet

SUMMARY:
To assess whether a rivaroxaban-based anticoagulation strategy, following successful TAVR, compared to an antiplatelet-based strategy, is superior in reducing death or first thromboembolic events (DTE).

To assess the primary bleeding events (PBE) of the rivaroxaban-based strategy compared to an antiplatelet-based strategy, following TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Successful TAVR (Transcatheter Aortic Valve Replacement) of an aortic valve stenosis (either native or valve-in-valve)

  * By iliofemoral or subclavian access
  * With any approved/marketed device

Exclusion Criteria:

* Atrial fibrillation (AF), current or previous, with an ongoing indication for oral anticoagulant treatment
* Any other indication for continued treatment with any oral anticoagulant (OAC)
* Known bleeding diathesis (such as but not limited to active internal bleeding, clinically significant bleeding, platelet count ≤ 50,000/mm3 at screening, hemoglobin level < 8.5 g/dL, active peptic ulcer or known gastrointestinal (GI) bleeding, history of intracranial hemorrhage or subdural hematoma)
* Any ongoing absolute indication for dual antiplatelet therapy (DAPT) at time of screening that is unrelated to the TAVR procedure
* Clinically overt stroke within the last 3 months
* Planned coronary or vascular intervention or major surgery
* Severe renal impairment (eGFR < 30 mL/min/1.73 m2) or on dialysis, or post-TAVR unresolved acute kidney injury with renal dysfunction stage 2 or higher
* Moderate and severe hepatic impairment (Child-Pugh Class B or C) or any hepatic disease associated with coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1653 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (123):
- United States (30):
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Evanston, Illinois
  - West Des Moines, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Morristown, New Jersey
  - Manhasset, New York
  - New York, New York
  - Roslyn, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Houston, Texas
  - Plano, Texas
  - Temple, Texas
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Falls Church, Virginia
  - Tacoma, Washington
- Austria (5):
  - Graz, Styria
  - Linz, Upper Austria
  - Wels, Upper Austria
  - Salzburg
  - Vienna
- Belgium (3):
  - Genk
  - Hasselt
  - Liège
- Canada (8):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Newmarket, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (2):
  - Brno
  - Prague
- Denmark (3):
  - Aarhus N
  - Copenhagen
  - Odense C
- France (6):
  - Angers
  - Brest
  - Chambray-lès-Tours
  - Lille
  - Paris
  - Toulouse
- Germany (31):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Konstanz, Baden-Wurttemberg
  - Lahr, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - Bad Neustadt an der Saale, Bavaria
  - Erlangen, Bavaria
  - München, Bavaria
  - Regensburg, Bavaria
  - Bad Nauheim, Hesse
  - Frankfurt am Main, Hesse
  - Fulda, Hesse
  - Rotenburg A.d. Fulda, Hesse
  - Hanover, Lower Saxony
  - Aachen, North Rhine-Westphalia
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Dortmund, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Krefeld, North Rhine-Westphalia
  - Neuss, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Leipzig, Saxony
  - Magdeburg, Saxony-Anhalt
  - Bad Segeberg, Schleswig-Holstein
  - Kiel, Schleswig-Holstein
  - Bad Berka, Thuringia
  - Berlin
  - Bremen
  - Hamburg
- Italy (5):
  - Bergamo, Lombardy
  - Milan, Lombardy
  - Catania, Sicily
  - Pisa, Tuscany
  - Padua, Veneto
- Netherlands (3):
  - Amsterdam
  - Breda
  - Rotterdam
- Norway (3):
  - Bergen
  - Oslo
  - Tromsø
- Poland (2):
  - Bielsko-Biala
  - Warsaw
- Seoul, South Korea
- Spain (5):
  - L'Hospitalet de Llobregat, Barcelona
  - Oviedo, Principality of Asturias
  - Barcelona
  - Madrid
  - Málaga
- Uppsala, Sweden
- Switzerland (5):
  - Basel, Canton of Basel-City
  - Lugano, Canton Ticino
  - Bern
  - Lucerne
  - Zurich
- United Kingdom (10):
  - Brighton, East Sussex
  - Southampton, Hampshire
  - Blackpool, Lancashire
  - Leicester, Leicestershire
  - Belfast, North Ireland
  - Newcastle upon Tyne, Tyne and Wear
  - Leeds, West Yorkshire
  - Edinburgh
  - London
  - Oxford

REFERENCES:
- [Derived] Okuno T, Dangas GD, Hengstenberg C, Sartori S, Herrmann HC, de Winter R, Gilard M, Tchetche D, Mollmann H, Makkar RR, Baldus S, De Backer O, Bendz B, Kini A, von Lewinski D, Mack M, Moreno R, Schafer U, Wohrle J, Seeger J, Snyder C, Nicolas J, Tijssen JGP, Welsh RC, Vranckx P, Valgimigli M, Mehran R, Kapadia S, Sondergaard L, Windecker S. Two-year clinical outcomes after successful transcatheter aortic valve implantation with balloon-expandable versus self-expanding valves: A subanalysis of the GALILEO trial. Catheter Cardiovasc Interv. 2022 Oct;100(4):636-645. doi: 10.1002/ccd.30370. Epub 2022 Aug 30. PMID 36040717
- [Derived] Wohrle J, Gilard M, Didier R, Kini A, Tavenier AH, Tijssen JGP, Sartori S, Snyder C, Nicolas J, Seeger J, Landmesser U, Tarantini G, Asgar A, Mollmann H, Thiele H, Capranzano P, Reimers B, Stefanini G, Moreno R, Petronio AS, Mikhail G, Kapadia S, Hildick-Smith D, Hengstenberg C, Mehran R, Windecker S, Dangas GD; GALILEO Investigator. Outcomes After Transcatheter Aortic Valve Implantation in Men Versus Women. Am J Cardiol. 2022 Oct 1;180:108-115. doi: 10.1016/j.amjcard.2022.06.035. Epub 2022 Aug 4. PMID 35934563
- [Derived] Dangas GD, Tijssen JGP, Wohrle J, Sondergaard L, Gilard M, Mollmann H, Makkar RR, Herrmann HC, Giustino G, Baldus S, De Backer O, Guimaraes AHC, Gullestad L, Kini A, von Lewinski D, Mack M, Moreno R, Schafer U, Seeger J, Tchetche D, Thomitzek K, Valgimigli M, Vranckx P, Welsh RC, Wildgoose P, Volkl AA, Zazula A, van Amsterdam RGM, Mehran R, Windecker S; GALILEO Investigators. A Controlled Trial of Rivaroxaban after Transcatheter Aortic-Valve Replacement. N Engl J Med. 2020 Jan 9;382(2):120-129. doi: 10.1056/NEJMoa1911425. Epub 2019 Nov 16. PMID 31733180
- [Derived] Piayda K, Zeus T, Sievert H, Kelm M, Polzin A. Subclinical leaflet thrombosis. Lancet. 2018 Mar 10;391(10124):937-938. doi: 10.1016/S0140-6736(18)30534-8. No abstract available. PMID 29536857
- [Derived] Windecker S, Tijssen J, Giustino G, Guimaraes AH, Mehran R, Valgimigli M, Vranckx P, Welsh RC, Baber U, van Es GA, Wildgoose P, Volkl AA, Zazula A, Thomitzek K, Hemmrich M, Dangas GD. Trial design: Rivaroxaban for the prevention of major cardiovascular events after transcatheter aortic valve replacement: Rationale and design of the GALILEO study. Am Heart J. 2017 Feb;184:81-87. doi: 10.1016/j.ahj.2016.10.017. Epub 2016 Oct 31. PMID 27892890
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 136 centers world-wide between 16 Dec 2015 (first patient's first visit) and 27 Nov 2018 (last patient's last visit).
Pre-assignment Details: A total of 1674 subjects were screened, of which 1644 were randomly assigned to either of the two treatment arms and 1608 subjects started treatment with study medication.
Groups:
- Rivaroxaban (Xarelto, BAY59-7939): Subjects were treated with Rivaroxaban (10mg once-daily) and ASA (Acetylsalicylic Acid) (75-100mg once-daily) within first 90 days after randomization. After 90 days, ASA was discontinued and rivaroxaban (10mg once-daily) was to be continued alone. In the event of NOAF (New Onset of Atrial Fibrillation), subjects should be switched to rivaroxaban (20/15mg once-daily) and ASA (75-100mg once-daily) within first 90 days. After 90 days, ASA was discontinued and rivaroxaban (20/15mg once-daily) was to be continued alone.
- Antiplatelet: Subjects were treated with clopidogrel (75mg once-daily) and ASA (75-100mg once-daily) within first 90 days after randomization. After 90 days, clopidogrel was discontinued and ASA (75-100mg once-daily) was to be continued alone. In the event of NOAF, subjects should start treatment of open-label VKA (Vitamin K antagonist) to target INR (international normalized ratio) 2 to 3 (according to guidelines) and ASA (75-100mg once-daily) within first 90 days. After 90 days, ASA was discontinued and VKA was to be continued alone.
Period: Overall Study
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Antiplatelet
Started | 826 | 818
Received Treatment | 801 | 807
Completed (Completed study procedures) | 799 | 792
Not Completed | 27 | 26
Not completed — Withdrawal by Subject | 21 | 21
Not completed — Lost to Follow-up | 5 | 5
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Antiplatelet | Total
Number analyzed (Participants) | 826 | 818 | 1644
Age, Continuous [Mean (Standard Deviation); unit: Years] | 80.38 (7.12) | 80.77 (5.99) | 80.57 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 400 | 413 | 813
  Male | 426 | 405 | 831
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 17 | 43
  Not Hispanic or Latino | 677 | 694 | 1371
  Unknown or Not Reported | 123 | 107 | 230
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 9 | 7 | 16
  White | 692 | 693 | 1385
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 123 | 115 | 238

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death or First Thromboembolic Event (DTE)
Description: Death or first adjudicated thromboembolic event (DTE), defined as composite of all-cause death, any stroke, myocardial infarction (MI), symptomatic valve thrombosis, pulmonary embolism (PE), deep vein thrombosis (DVT), and non-central nervous system (CNS) systemic embolism.
Time Frame: Through study completion, on average 14 months
Population: Safety analysis set (SAF): Included all randomized subjects who had been exposed to study drug at least once (1608 subjects overall).
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Antiplatelet
Number analyzed (Participants) | 801 | 807
Participants | 68 | 63
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Antiplatelet; H0: HR(t)>=1.20 for all time points t>=0, (i.e. "the hazard for the primary efficacy endpoint in the rivaroxaban-based treatment group is more than 20% larger than that in the antiplatelet-based control group"); Test type: Non-Inferiority — 1-sided Confidence interval; Hazard Ratio (HR) = 1.2089302, 97.5% CI 1-sided [upper limit 1.7040824]

2. Primary Outcome: Number of Participants With Death or First Thromboembolic Event (DTE)
Description: as for outcome 1
Time Frame: Through study completion, on average 16 months
Population: Full analysis set (FAS): Included all randomized subjects and results presented according to randomized treatment arm (1644 subjects overall)
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Antiplatelet
Number analyzed (Participants) | 826 | 818
Participants | 105 | 78
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Antiplatelet; Test type: Superiority — 2-sided Log Rank test; p = 0.04223, Log Rank; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [1.01 to 1.81]

3. Primary Outcome: Number of Participants With Primary Bleeding Event (PBE)
Description: PBE is defined according to VARC (Valve Academic Research Consortium) definitions as the adjudicated composite of: Life-threatening, disabling or major bleeding.
Time Frame: Through study completion, on average 16 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Antiplatelet
Number analyzed (Participants) | 826 | 818
Participants | 46 | 31
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Antiplatelet; Test type: Other — Descriptive. 2-sided Log Rank test; p = 0.07745, Log Rank; Hazard Ratio (HR) = 1.50, 95% CI 2-sided [0.95 to 2.37] — Estimates for HRs are based on Cox proportional hazards model. HRs >1 indicate a higher hazard rate in the rivaroxaban arm compared with the antiplatelet arm

4. Secondary Outcome: Number of Participants With Net-clinical Benefit
Description: The net-clinical-benefit defined as the adjudicated composite of all-cause death, any stroke, myocardial infarction, symptomatic valve thrombosis, pulmonary embolism, deep vein thrombosis, non-CNS systemic embolism (efficacy); VARC life-threatening, disabling and VARC major bleeds (safety).
Time Frame: Through study completion, on average 16 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Antiplatelet
Number analyzed (Participants) | 826 | 818
Participants | 137 | 100
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Antiplatelet; Test type: Superiority — 2-sided Log Rank test; p = 0.01156, Log Rank; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [1.08 to 1.80] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Number of Participants With Cardiovascular Death or Thromboembolic Event
Description: Composite of CV-death, any stroke, myocardial infarction (MI), symptomatic valve thrombosis, pulmonary embolism (PE), deep vein thrombosis (DVT), and non-central nervous system (CNS) systemic embolism (per adjudication).
Time Frame: Through study completion, on average 16 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Antiplatelet
Number analyzed (Participants) | 826 | 818
Participants | 83 | 68
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Antiplatelet; Test type: Superiority — 2-sided Log Rank test; p = 0.21595, Log Rank; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.89 to 1.69] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Number of Participants With TIMI (Thrombolysis In Myocardial Infarction) Major / Minor Bleeds
Description: Composite of TIMI major and minor bleedings
Time Frame: Through study completion, on average 16 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Antiplatelet
Number analyzed (Participants) | 826 | 818
Participants | 42 | 24
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Antiplatelet; Test type: Other — Descriptive. 2-sided Log Rank test; p = 0.02216, Log Rank; Hazard Ratio (HR) = 1.78, 95% CI 2-sided [1.08 to 2.94] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Number of Participants With ISTH (International Society on Thrombosis and Haemostasis) Major Bleeds
Description: ISTH major bleeds
Time Frame: Through study completion, on average 16 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Antiplatelet
Number analyzed (Participants) | 826 | 818
Participants | 49 | 30
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Antiplatelet; Test type: Other — Descriptive. 2-sided Log Rank test; p = 0.02702, Log Rank; Hazard Ratio (HR) = 1.66, 95% CI 2-sided [1.05 to 2.62] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Number of Participants With Composite Bleeding Endpoint of BARC (Bleeding Academic Research Consortium) 2, 3, or 5 Bleeds
Description: Composite of BARC 2,3 or 5 bleedings
Time Frame: Through study completion, on average 16 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Antiplatelet
Number analyzed (Participants) | 826 | 818
Participants | 148 | 85
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Antiplatelet; Test type: Other — Descriptive. 2-sided Log Rank test; p = 0.00001, Log Rank; Hazard Ratio (HR) = 1.84, 95% CI 2-sided [1.41 to 2.41] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Through study completion, on average 14 months. Timeframe for All-Cause Mortality: After study medication start until last contact date.
Groups:
- Rivaroxaban Arm: Subjects were treated with Rivaroxaban (10mg once-daily) and ASA (75-100mg once-daily) within first 90 days after randomization. After 90 days, ASA was discontinued and rivaroxaban (10mg once-daily) was to be continued alone. In the event of NOAF (New Onset of Atrial Fibrillation), subjects should be switched to rivaroxaban (20/15mg once-daily) and ASA (75-100mg once-daily) within first 90 days. After 90 days, ASA was discontinued and rivaroxaban (20/15mg once-daily) was to be continued alone.
- Antiplatelet Arm: Subjects were treated with clopidogrel (75mg once-daily) and ASA (75-100mg once-daily) within first 90 days after randomization. After 90 days, clopidogrel was discontinued and ASA (75-100mg once-daily) was to be continued alone. In the event of NOAF, subjects should start treatment of open-label VKA (Vitamin K antagonist) to target INR (international normalized ratio) 2 to 3 (according to guidelines) and ASA (75-100mg once-daily) within first 90 days. After 90 days, ASA was discontinued and VKA was to be continued alone.
Arm/Group | Rivaroxaban Arm | Antiplatelet Arm
All-Cause Mortality (participants affected / at risk) | 70/801 | 43/807
Serious Adverse Events (participants affected / at risk) | 296/801 | 282/807
Other Adverse Events (participants affected / at risk) | 359/801 | 302/807
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban Arm (N=801) | Antiplatelet Arm (N=807)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 17 (19) | 25 (27)
Atrial flutter (Cardiac disorders) | 4 (4) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 12 (12) | 15 (15)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 3 (3)
Atrioventricular block second degree (Cardiac disorders) | 4 (4) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Bundle branch block left (Cardiac disorders) | 4 (4) | 6 (6)
Cardiac arrest (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac failure (Cardiac disorders) | 16 (19) | 16 (22)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 5 (10)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 8 (8) | 3 (4)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 2 (2) | 2 (2)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 5 (8) | 3 (5)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0)
Trifascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 4 (4)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 2 (2)
Neuroacanthocytosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Primary adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (4)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Macular detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coeliac artery stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 5 (5) | 5 (5)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 2 (2)
Sudden cardiac death (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 1 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Pacemaker generated arrhythmia (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 3 (4) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 2 (3) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 4 (4)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 8 (8) | 7 (7)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 2 (3)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 23 (28) | 22 (23)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 7 (7) | 3 (3)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 4 (4) | 1 (1)
Groin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (5) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound abscess (Infections and infestations) | 0 (0) | 1 (1)
Renal cyst infection (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 3 (3)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Cardiac valve abscess (Infections and infestations) | 1 (1) | 0 (0)
Dermo-hypodermitis (Infections and infestations) | 1 (2) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Septic encephalopathy (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Medical device site joint infection (Infections and infestations) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 12 (12) | 5 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pancreatic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial bypass stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural hypoparathyroidism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Product administration error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Inflammatory marker increased (Investigations) | 1 (1) | 0 (0)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
Transvalvular pressure gradient increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 2 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (4)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Axonal neuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 9 (9) | 4 (4)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (3) | 1 (2)
Extrapyramidal disorder (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 1 (1)
Hypotonia (Nervous system disorders) | 2 (2) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 0 (0)
Sciatica (Nervous system disorders) | 4 (6) | 2 (2)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 19 (20) | 23 (25)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (2)
Ballismus (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (3) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (3) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1)
Panic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 10 (10) | 17 (17)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cochlea implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 3 (3)
Incisional hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 3 (3) | 0 (0)
Skin cyst excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Dental operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Ear operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Eyelid operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker adjustment (Surgical and medical procedures) | 0 (0) | 1 (1)
Transcatheter arterial chemoembolisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 5 (5)
Hypertensive crisis (Vascular disorders) | 3 (3) | 5 (6)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 8 (8)
Undersensing (Product Issues) | 0 (0) | 1 (1)
Device battery issue (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban Arm (N=801) | Antiplatelet Arm (N=807)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 43 (44) | 44 (45)
Atrial flutter (Cardiac disorders) | 2 (2) | 5 (5)
Atrial tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 7 (7) | 8 (8)
Bradycardia (Cardiac disorders) | 3 (3) | 2 (2)
Bundle branch block left (Cardiac disorders) | 6 (6) | 7 (7)
Cardiac failure (Cardiac disorders) | 14 (15) | 11 (11)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 3 (3)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 7 (7) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 17 (17) | 8 (8)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (3) | 7 (7)
Cataract (Eye disorders) | 2 (2) | 5 (6)
Lacrimation increased (Eye disorders) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 3 (3) | 2 (2)
Visual impairment (Eye disorders) | 6 (6) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 8 (8) | 6 (6)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 9 (11)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 10 (10) | 4 (4)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Asthenia (General disorders) | 4 (4) | 2 (2)
Chest pain (General disorders) | 10 (10) | 12 (12)
Fatigue (General disorders) | 13 (15) | 7 (7)
Gait disturbance (General disorders) | 2 (2) | 2 (2)
Oedema (General disorders) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 16 (16) | 20 (21)
Pyrexia (General disorders) | 1 (1) | 2 (4)
Peripheral swelling (General disorders) | 0 (0) | 3 (3)
General physical health deterioration (General disorders) | 0 (0) | 3 (3)
Drug intolerance (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 5 (5)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 9 (10) | 12 (12)
Cellulitis (Infections and infestations) | 1 (1) | 4 (4)
Conjunctivitis (Infections and infestations) | 2 (2) | 2 (2)
Cystitis (Infections and infestations) | 3 (3) | 3 (3)
Erysipelas (Infections and infestations) | 1 (1) | 2 (2)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 2 (2)
Gingivitis (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 2 (2)
Infection (Infections and infestations) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (5)
Oesophageal candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 5 (6) | 10 (10)
Pulpitis dental (Infections and infestations) | 4 (4) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 30 (33) | 19 (21)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 18 (18) | 16 (16)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 11 (11) | 8 (11)
Skin laceration (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 4 (4)
Blood glucose increased (Investigations) | 3 (3) | 0 (0)
Blood pressure increased (Investigations) | 4 (4) | 4 (4)
C-reactive protein increased (Investigations) | 1 (1) | 3 (3)
Electrocardiogram QRS complex prolonged (Investigations) | 2 (2) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 3 (3)
International normalised ratio abnormal (Investigations) | 0 (0) | 3 (3)
Intraocular pressure increased (Investigations) | 0 (0) | 2 (2)
Weight increased (Investigations) | 0 (0) | 2 (2)
Ejection fraction decreased (Investigations) | 2 (2) | 5 (5)
Transvalvular pressure gradient increased (Investigations) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Gout (Metabolism and nutrition disorders) | 7 (8) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 5 (6)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 2 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (3) | 1 (1)
Dementia (Nervous system disorders) | 4 (4) | 2 (2)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 32 (32) | 16 (16)
Headache (Nervous system disorders) | 10 (10) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 3 (3)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 5 (5) | 3 (3)
Sciatica (Nervous system disorders) | 3 (3) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 10 (10) | 15 (16)
Cognitive disorder (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 2 (2)
Nocturia (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (2)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 4 (4) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 8 (8)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 6 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (5)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 10 (10) | 0 (0)
Cataract operation (Surgical and medical procedures) | 6 (9) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 3 (3) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 26 (26) | 28 (28)
Hypertensive crisis (Vascular disorders) | 4 (4) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 10 (11)
Intermittent claudication (Vascular disorders) | 2 (2) | 1 (1)
Lymphoedema (Vascular disorders) | 4 (4) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (6) | 2 (2)
Peripheral venous disease (Vascular disorders) | 0 (0) | 2 (2)
Device dislocation (Product Issues) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-08-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT02556203/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT02556203/SAP_001.pdf